CLINICAL TRIAL: NCT01691430
Title: A Randomized, Controlled Trial of Cranberry Capsules for UTI Prevention in Nursing Home Residents
Brief Title: A Trial of Cranberry Capsules for Urinary Tract Infection Prevention in Nursing Home Residents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1112009472; 2P30AG021342-11 (NIH); 1R01AG041153-01A1 (NIH)
Record Dates: First submitted 2012-08-09; First posted 2012-09-24 (Estimated); Results first posted 2018-01-29 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Bacteriuria
MeSH Terms: conditions — Bacteriuria

STUDY DESIGN:
Intervention Model Description: Participants were randomized to cranberry or placebo capsules.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 cranberry capsules (Active Comparator): Experimental: 2 cranberry capsules
  Interventions: Dietary Supplement: 2 cranberry capsules
- 2 placebo capsules (Placebo Comparator): Experimental: 2 placebo capsules qd
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 2 cranberry capsules — Two cranberry capsules qd (each capsule containing 36mg proanthocyanidin, total 72mg PAC)
  Arms: 2 cranberry capsules
Dietary Supplement: Placebo — Two placebo capsules qd (each capsule containing 36mg proanthocyanidin, total 72mg PAC)
  Arms: 2 placebo capsules

SUMMARY:
Urinary tract infection (UTI) is the most common infection in nursing home residents, and bacteriuria is the greatest trigger for antimicrobial therapy in the nursing home setting. The primary aim of this study is to test the efficacy of two oral cranberry capsules per day in the reduction of bacteriuria plus pyuria in female nursing home residents. These aims will be accomplished by conducting a double blind randomized placebo controlled efficacy trial of two oral cranberry capsules daily versus placebo in a cohort of Connecticut female nursing home residents.

ELIGIBILITY:
Inclusion Criteria:

1. female residents;
2. long term residents
3. English speaking; and
4. age ≥ 65 years.

Exclusion Criteria:

1. residents that are not expected to be in the nursing home for at least one month (i.e., short term rehabilitation, pending discharge, terminal [life expectancy < 1 month]);
2. residents who are on chronic suppressive antibiotic or anti-infective (i.e., mandelamine) therapy for recurrent UTI;
3. residents with end stage renal disease on dialysis (they do not regularly produce urine);
4. residents unable to produce a baseline clean catch urine specimen for collection;
5. residents on warfarin therapy because of a potential interaction of warfarin and cranberry juice;
6. residents with a history of nephrolithiasis because cranberry may increase the risk of nephrolithiasis;
7. have an indwelling bladder catheter in place;
8. have an allergy to cranberry products;
9. are being treated with cranberry products;
10. residence <4 weeks.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 185 (Actual)
Dates: Start 2012-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Juthani-Mehta, M.D., Principal Investigator — Yale University
Locations (21):
- United States (21):
  - Branford Hills Health Care, Branford, Connecticut
  - Northbridge Health Care Center, Bridgeport, Connecticut
  - Bridgeport Health Care Center, Bridgeport, Connecticut
  - Bridgeport Manor, Bridgeport, Connecticut
  - Riverside Health & Rehabilitation Center, East Hartford, Connecticut
  - Ludlowe Health Care Center, Fairfield, Connecticut
  - Glastonbury Health Care Center, Glastonbury, Connecticut
  - The Nathaniel Witherell, Greenwich, Connecticut
  - Arden House Care and Rehabilitation Center, Hamden, Connecticut
  - Hamden Health Care Center, Hamden, Connecticut
  - Avery Heights, Hartford, Connecticut
  - Wadsworth Glen Health Care and Rehabilitation Center, Middletown, Connecticut
  - Water's Edge Center for Health & Rehabilitation, Middletown, Connecticut
  - Grimes Center, New Haven, Connecticut
  - Mary Wade Home, New Haven, Connecticut
  - Advanced Nursing & Rehab Center of New Haven, New Haven, Connecticut
  - Shady Knoll Health Center, Seymour, Connecticut
  - Lord Chamberlain Nursing & Rehabilitation Center, Stratford, Connecticut
  - Village Green of Wallingford, Wallingford, Connecticut
  - Abbott Terrace Health Center, Waterbury, Connecticut
  - Hughes Health & Rehab Center, West Hartford, Connecticut

REFERENCES:
- [Derived] Williams G, Stothart CI, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Nov 10;11(11):CD001321. doi: 10.1002/14651858.CD001321.pub7. PMID 37947276
- [Derived] Williams G, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Apr 17;4(4):CD001321. doi: 10.1002/14651858.CD001321.pub6. PMID 37068952
- [Derived] Datta R, Trentalange M, Van Ness PH, McGloin JM, Guralnik JM, Miller ME, Walkup MP, Nadkarni N, Pahor M, Gill TM, Quagliarello V, Juthani-Mehta M; LIFE Study Group. Serious adverse events of older adults in nursing home and community intervention trials. Contemp Clin Trials Commun. 2017 Dec 21;9:77-80. doi: 10.1016/j.conctc.2017.12.004. eCollection 2018 Mar. PMID 29696228
- [Derived] Juthani-Mehta M, Van Ness PH, Bianco L, Rink A, Rubeck S, Ginter S, Argraves S, Charpentier P, Acampora D, Trentalange M, Quagliarello V, Peduzzi P. Effect of Cranberry Capsules on Bacteriuria Plus Pyuria Among Older Women in Nursing Homes: A Randomized Clinical Trial. JAMA. 2016 Nov 8;316(18):1879-1887. doi: 10.1001/jama.2016.16141. PMID 27787564

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from nursing homes within 50 miles of New Haven.
Pre-assignment Details: 806 patients were eligible, 558 declined to participate. Of the 248 consented, 63 were found to be ineligible after consent, leaving 185 to randomize.
Period: Overall Study
Arm/Group | 2 Cranberry Capsules | 2 Placebo Capsules
Started | 92 | 93
Received Medication | 92 | 93
Completed | 70 | 73
Not Completed | 22 | 20
Not completed — Death | 17 | 16
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Population: Inclusion criteria were (1) female; (2) long-term care residents; (3) English speaking; and (4) 65 years or older.
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 Cranberry Capsules | 2 Placebo Capsules | Total
Number analyzed (Participants) | 92 | 93 | 185
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 92 | 93 | 185
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 93 | 185
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 83 | 84 | 167
  Non-White | 9 | 9 | 18
Bacteriuria plus pyuria [Number; unit: participants] | 27 | 32 | 59

OUTCOME MEASURES:

1. Primary Outcome: Participants With Urine Cultures With Bacteriuria (>100,000 Cfu/ml or >=100,000 Cfu/ml) Plus Pyuria (Any WBC)
Description: Clean catch urine cultures and urinalyses will be obtained every two months for each participant for study purposes.
Time Frame: One year
Population: 147 subjects completed 1 year, 33 died. 20 subjects, 9 in the treatment group v 11 in the control group, became incontinent prior to the first time point, thus unable to provide any urine. 45 subjects stopped taking the capsules, 24 in treatment and 21 in control; 21 refused, 19 transitioned to hospice, 4 started warfarin, and 1 refused via family.
Measure: Number; unit: participants
Arm/Group | 2 Cranberry Capsules | 2 Placebo Capsules
Number analyzed (Participants) | 92 | 93
participants
  Baseline | 26 | 32
  2 months: number analyzed (Participants) | 76 | 78
  2 months | 21 | 27
  4 months: number analyzed (Participants) | 63 | 65
  4 months | 15 | 26
  6 months: number analyzed (Participants) | 64 | 67
  6 months | 13 | 20
  8 months: number analyzed (Participants) | 55 | 60
  8 months | 14 | 14
  10 months: number analyzed (Participants) | 51 | 54
  10 months | 15 | 13
  12 months: number analyzed (Participants) | 44 | 46
  12 months | 12 | 9

2. Secondary Outcome: Number of Episodes of Symptomatic UTI
Description: Suspected UTI episodes that are recorded in the medical record by the primary provider will be reviewed by chart review, symptoms will be recorded, and two adjudicators will determine if the definition of symptomatic UTI is met.
Time Frame: One year
Measure: Number; unit: symptomatic urinary tract infections
Arm/Group | 2 Cranberry Capsules | 2 Placebo Capsules
Number analyzed (Participants) | 92 | 93
symptomatic urinary tract infections | 10 | 12

3. Secondary Outcome: Number of Hospitalizations
Time Frame: One year
Measure: Number; unit: hospitilizations
Arm/Group | 2 Cranberry Capsules | 2 Placebo Capsules
Number analyzed (Participants) | 92 | 93
hospitilizations | 33 | 50

4. Secondary Outcome: Number of Deaths
Time Frame: One year
Measure: Number; unit: participants
Arm/Group | 2 Cranberry Capsules | 2 Placebo Capsules
Number analyzed (Participants) | 92 | 93
participants | 17 | 16

5. Secondary Outcome: Number of Antibiotic Prescriptions
Description: Chart review will be performed to determine the names and duration of antibiotic prescriptions prescribed by the primary provider on each participant.
Time Frame: One year
Measure: Number; unit: prescriptions
Arm/Group | 2 Cranberry Capsules | 2 Placebo Capsules
Number analyzed (Participants) | 92 | 93
prescriptions | 1415 | 1883

6. Secondary Outcome: Bacteriuria With Multidrug-resistant Gram-negative Bacilli
Description: All urine culture data will be reviewed to determine presence of multidrug-resistant gram-negative bacilli (resistance to ≥3 of the following antibiotics: ampicillinsulbactam,cefazolin, ceftriaxone, ceftazidime, fluoroquinolones, piperacillin-tazobactam, meropenem, imipenem, and trimethoprim-sulfamethoxazole).
Time Frame: One year
Measure: Number; unit: episodes
Arm/Group | 2 Cranberry Capsules | 2 Placebo Capsules
Number analyzed (Participants) | 92 | 93
episodes | 9 | 24

7. Secondary Outcome: Number of Antibiotic Prescriptions for Suspected UTI
Description: Chart review will be performed to determine the names and duration of antibiotic prescriptions prescribed by the primary provider on each participant's suspected UTI.
Time Frame: One Year
Measure: Number; unit: prescriptions
Arm/Group | 2 Cranberry Capsules | 2 Placebo Capsules
Number analyzed (Participants) | 92 | 93
prescriptions | 692 | 909

8. Other Pre Specified Outcome: Number of Adverse Events in Participants
Time Frame: One year
Measure: Number; unit: adverse events
Arm/Group | 2 Cranberry Capsules | 2 Placebo Capsules
Number analyzed (Participants) | 92 | 93
adverse events
  Serious unrelated | 50 | 66
  non-serious unrelated | 1731 | 1966
  non-serious related | 7 | 7

9. Other Pre Specified Outcome: Adherence to Capsule Intake by All Participants
Description: measured by capsules removed from blister packs
Time Frame: One year
Measure: Number; unit: percentage of capsules
Arm/Group | 2 Cranberry Capsules | 2 Placebo Capsules
Number analyzed (Participants) | 92 | 93
percentage of capsules | 77.5 | 82.6

10. Secondary Outcome: Subjects With 1, 2, or 3 Episodes of UTIs
Description: as for outcome 2
Time Frame: One year
Population: There were 10 symptomatic UTIs in the treatment group (8 participants with 1 episode and 1 participant with 2 episodes) and 12 symptomatic UTIs in the control group (7 participants with 1 episode, 1 participant with 2 episodes, and 1 participant with 3 episodes).
Measure: Number; unit: participants
Arm/Group | 2 Cranberry Capsules | 2 Placebo Capsules
Number analyzed (Participants) | 92 | 93
participants
  1 episode | 8 | 7
  2 episodes | 1 | 1
  3 episodes | 0 | 1

ADVERSE EVENTS:
Arm/Group | 2 Cranberry Capsules | 2 Placebo Capsules
Serious Adverse Events (participants affected / at risk) | 50/92 | 66/93
Other Adverse Events (participants affected / at risk) | 92/92 | 93/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 Cranberry Capsules (N=92) | 2 Placebo Capsules (N=93)
Hospitalization (General disorders) | 33 | 50
Death (General disorders) | 17 (17) | 16 (16)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2 Cranberry Capsules (N=92) | 2 Placebo Capsules (N=93)
Abnormal blood glucose (Blood and lymphatic system disorders) | 9 | 11
Acute chest pain (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Acute renal failure (Renal and urinary disorders) | 1 | 0
Altered mental status (Psychiatric disorders) | 53 | 61
Anemia (Blood and lymphatic system disorders) | 4 | 4
Back Pain (General disorders) | 11 | 17
Blood pressure alteration (Blood and lymphatic system disorders) | 14 | 14
constipation (Gastrointestinal disorders) | 47 | 51
dehydration (General disorders) | 1 | 1
dizziness (Nervous system disorders) | 4 | 6
ear problem (Ear and labyrinth disorders) | 6 | 11
edema (General disorders) | 17 | 21
exposure to influenza (Infections and infestations) | 10 | 13
eye infection (Eye disorders) | 18 | 17
Fall (General disorders) | 48 | 55
fever (General disorders) | 18 | 21
GI disturbance (Gastrointestinal disorders) | 53 | 53
Generalized malaise (General disorders) | 29 | 27
headache (General disorders) | 10 | 19
insomnia (General disorders) | 6 | 10
joint pain (General disorders) | 36 | 31
lab abnormality (General disorders) | 42 | 43
leg pain (Musculoskeletal and connective tissue disorders) | 8 | 9
oral cavity disturbance (General disorders) | 34 | 25
respiratory difficulty (Respiratory, thoracic and mediastinal disorders) | 55 | 59
skin/soft tissue event (Skin and subcutaneous tissue disorders) | 71 | 83
Urinary Tract Infection (Renal and urinary disorders) | 33 | 44
weight gain (Metabolism and nutrition disorders) | 42 | 48
weight loss (Metabolism and nutrition disorders) | 62 | 74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No